CLINICAL TRIAL: NCT01710371
Title: Quantitative PET Imaging of Pancreatic Beta-Cell Mass in Healthy Overweight/Obese Subjects, Subjects With Prediabetes, and Type 2 Diabetes Patients With 18F-FP-DTBZ (18F-AV-133)
Brief Title: Quantitative 18F-AV-133 PET Imaging in Subjects With Diabetes and Healthy Controls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A9001458
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — florbenazine F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arginine Stimulation Testing (Experimental): Establish the methodology for glucose enhanced arginine stimulation testing (AST).
  Interventions: Drug: 10% Arginine Hydrochloride-R-Gene 10
- PET Imaging (Experimental): Determine if pancreatic PET-determined binding measures of 18F-AV-133 differ in up to 60 subjects determined to be at one of four stages of the natural history of Type 2 Diabetes: Healthy Overweight/obese Volunteers (HOV), Subjects with Pre-diabetes (PD) and Type 2 Diabetes mellitus (T2DM).
  Interventions: Drug: 18F-AV-133; Drug: 10% Arginine Hydrochloride-R-Gene 10

INTERVENTIONS:
Drug: 18F-AV-133 — 296 MBq (8 mCi)
  Arms: PET Imaging
Drug: 10% Arginine Hydrochloride-R-Gene 10

SUMMARY:
To evaluate 18F-AV-133 imaging of the pancreas in patients with early type 2 diabetes, late type 2 diabetes, subjects with pre-diabetes and in healthy overweight/obese control subjects. These subjects will also be evaluated for beta-cell function as measured by the insulin and C-peptide response to a challenge with intravenous arginine under basal and glucose enhanced conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects of non-childbearing potential between the ages of 30 and 65 years inclusive.
* Able to tolerate PET, PET/CT and MR imaging
* Estimated creatinine clearance >= 60mL/min
* Informed consent documents signed and dated by subject
* Subjects must be willing and able to comply with all scheduled visits, treatments laboratory tests, scans and other study procedures.
* In addition, subjects must meet classification requirements for one of the following

  1. Healthy Overweight
  2. Pre-diabetes
  3. T2DM
* (T2DM only) Subjects with other chronic medical conditions (besides diabetes) that are well controlled and stable on medication are acceptable for inclusion in this study.

Exclusion Criteria:

* Subjects who are affiliated with or relatives of staff members of either the site or Pfizer directly involved in the conduct of the trial.
* Conditions which in the opinion of the study investigator may interfere with the subject's ability to participate in the study
* History of allergic reaction to drug/contrast agent or history of drug/alcohol abuse
* Subjects who have received investigational medications within the last 30 days or a radiopharmaceutical in the past 7 days.
* Pregnant or nursing females; females of childbearing potential.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Optimal PET-determined mean pancreatic Binding Potential of 18F-AV-133 | PET visit 1
Optimal PET-determined mean pancreatic Standardized Uptake Value (SUV) of 18F-AV-133 | PET visit 1
Optimal PET-determined mean pancreatic Volume of Distribution (VT) of 18F-AV-133 | PET visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, New Haven, Connecticut, United States